CLINICAL TRIAL: NCT00581282
Title: Brain Imaging Studies of the Effects of Cocaine Abstinence
Status: Withdrawn | Type: Observational
Why Stopped: Nonapplicable clinical trial
Sponsor: University of California, Irvine (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: HS#2004-4019
Record Dates: First submitted 2007-12-21; First posted 2007-12-27 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Substance Abuse Disorder
Keywords: Cocaine abstinence; PET scan
MeSH Terms: conditions — Substance-Related Disorders | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Cocaine abstinent group
  Interventions: Radiation: PET scan; Other: fMRI
- 2: Normal healthy control group
  Interventions: Radiation: PET scan; Other: fMRI

INTERVENTIONS:
Radiation: PET scan — positron emission tomography PET scan
Other: fMRI — functional magnetic resonance imaging fMRI

SUMMARY:
This study evaluates theories regarding cocaine abstinence which propose that increased presynaptic and postsynaptic dopamine activity and increased serotonin activity are associated with abstinence in cocaine dependent subjects at the beginning and three to six months after a treatment program. We are using positron emission tomography (PET), Magnetic Resonance Imaging (MRI) and diffusion tensor imaging (DTI) in cortical and subcortical areas in a series of brain imaging studies testing these theories of abnormalities in the dopamine and serotonin system for cocaine addiction by examining the distribution of 18F-fallypride, 18F-altanserin, and FDG. We are evaluating genetic theories associated with cocaine addiction through the examination of genetic markers and functional genomics.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria include:

1. Subjects must be male or female and English speaking.
2. Subjects must be adults with a history of diagnosis of cocaine dependence disorder (n=20) who are under supervised treatment for dependence or normal control (n=10).
3. Subjects must be between 21 to 65 years of age.

Exclusion Criteria:

Exclusion criteria include:

1. Suicidality or psychosis.
2. Head injury, kidney or bladder disease or any unstable or serious medical conditions.
3. Prior exposure to radiation (including diagnostic or treatment x-rays), which might cause subjects to exceed standard guidelines.
4. Unwillingness or inability to adhere to the requirements of the study.
5. Donation or large loss of blood (>400 ml) within the past month.
6. Current or very recent illnesses, painful conditions or other disorders, which in the judgment of the investigators, might invalidate the scientific goals of the study or pose undesirable difficulties or risks for subjects.
7. Pregnancy or breast feeding.
8. Individuals who would be unable to undergo a magnetic resonance imaging (MRI) scan, for example, individuals who suffer from claustrophobia, or who have metal clips in their body, metallic prostheses (i.e., replacement body parts, such as a hip joint), a pacemaker, or other pieces of metal in their body (shrapnel, metal filings, etc.).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in cocaine dependency treatment program Normal Healthy Control Subjects
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-12 (Actual); Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
PET scans, fMRI scans | The beginning and three to six months after a treatment program

CONTACTS AND LOCATIONS:
Overall Officials: Joseph C Wu, M.D., Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Brain Imaging Center, Irvine, California, United States